CLINICAL TRIAL: NCT06577909
Title: Prednisone Plus IVIg Compared With Prednisone for Immune Thrombocytopenia During Pregnancy
Brief Title: Prednisone Plus IVIg vs. Prednisone for ITP During Pregnancy
Acronym: IVIg
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-ITP023
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia; pregnancy; therapy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone; Lead; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combination group (Experimental): Prednisone 20mg per day×4 weeks and IVIg 400mg/kg per day（≤20g per day）×5 days
  Interventions: Drug: Prednisone; Drug: IVIg
- The prednisone group (Active Comparator): Prednisone 20mg per day×4 weeks
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone po, 20mg per day for 4 weeks, if response (Plt 30-100×100^g/L), gradually taper to the maintenance dose of 5-10mg per day until 6 weeks after delivery; if not response, gradually taper to withdrawal.
  Other Names: Pre
Drug: IVIg — IVIg 400mg/kg (≤20g for the total dose) per day for 5 days, and repeated in the case of lack of response by day 14
  Other Names: intravenous immunoglobulin
  Arms: The combination group

SUMMARY:
This is a prospective, randomized, open-label, multicenter clinical trial study to compare the efficacy and safety of prednisone plus IVIg to prednisone monotherapy in the treatment of immune thrombocytopenia (ITP) in pregnancy.

DETAILED DESCRIPTION:
The investigators are undertaking a prospective, parallel group, multicenter, randomized controlled trial in pregnant patients with treat-naive ITP. A total of 100 participants are randomized to two groups with the 1:1 ratio: prednisone plus IVIg group versus prednisone monotherapy group. Participants will receive prednisone 20mg per day for 4 weeks plus IVIg 400mg/Kg (total dose ≤20g per day) for 5 days or prednisone 20mg monotherapy per day for 4 weeks. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Time to response and platelet counts of newborns are investigated. Adverse events including participants and their newborns are also recorded throughout and after the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years old;
2. Meet the diagnostic criteria for immune thrombocytopenia;
3. Pregnant women with ITP without ITP-specific treatments during pregnancy;
4. Gestational weeks ≥12 weeks;
5. Platelet count <30×10^9/L, accompanied with or without bleeding symptoms.
6. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Have a known diagnosis of other autoimmune diseases, confirmed medical history or laboratory findings within positive anti-nuclear antibodies (>1:80), anti-cardiolipin antibodies, lupus anticoagulant factors or direct Coombs' test.
2. Thrombocytopenia caused by pregnancy-specific conditions, such as gestational thrombocytopenia, preeclampsia, the HELLP syndrome and acute fatty liver of pregnancy.
3. Secondary thrombocytopenia such as drug-related thrombocytopenia, vaccine-related thrombocytopenia, lymphoproliferative disorders, severe infection, hepatic cirrhosis and so on.
4. With other underlying diseases that may cause thrombocytopenia, such as: malignant disease, megaloblastic anemia, aplastic anemia, myelodysplasia syndrome, myeloid fibrosis, disseminated intravascular coagulation, thrombotic thrombocytopenic purpura, Hemolytic uremic syndrome, disseminated intravascular coagulation and so on;
5. Current HIV infection or hepatitis B virus or hepatitis C virus infections;
6. With severe heart, kidney, liver or respiratory dysfunction;
7. With the medical history of mental illness;
8. Have allergic reaction to prednisone or IVIg;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response | 4 weeks
  Achieving a platelet count of≥30×10^9/L and at least a doubling of the baseline platelet count without administration of any other ITP-specific treatment, and the absence of bleeding

SECONDARY OUTCOMES:
Complete Response | 4 weeks
  Platelet count ≥100×10^9/L measured on 2 occasions at least 7 days apart and the absence of bleeding
Early response | 1 week
  Platelet count ≥30×10^9/L and at least doubling baseline at 1 week
relapse | 1 year
  After the treatment is effective, the platelet count drops below 30×10^9/L or drops to less than 2 times the basal value, or bleeding symptoms occur
Time to Response | 4 weeks
  The day achieving OR
Time to relapse (duration of efficacy) | 1 year
  The time from achievement of CR or R to time of relapse
Platelet counts at delivery | At delivery
  Platelet counts at delivery
Platelet counts of newborns | up to 42 days per newborn
  Platelet counts of d1, 3, and 7 of newborns, extended to d42 if thrombocytopenia occurs
Adverse events in parturients | 2 years
  up to 2 years per subject

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, Professor, Principal Investigator — Peking University Insititute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China